CLINICAL TRIAL: NCT05625581
Title: Clinical Study on the Efficacy and Safety of Tofatib and Cyclophosphamide in the Treatment of Active IgG4 Related Diseases
Brief Title: Tofatib Treatment for IgG4-related Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CHEC2022-175
Record Dates: First submitted 2022-11-10; First posted 2022-11-23 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: IgG4-related Disease
MeSH Terms: conditions — Immunoglobulin G4-Related Disease | interventions — tofacitinib; Cyclophosphamide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — TB infection screening test, hepatitis B antibody, hepatitis C antibody, syphilis antibody, HIV antibody, tumor full set; Blood routine, liver and kidney function, blood lipid, blood sugar, coagulation function, urine routine; Blood sink, CRP, immunoglobulin, complement, IgG4, ANA profile, RF, ANCA, lymphocyte subsets, and cytokines
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Glucocorticosteroids combined with Cyclophosphamide Group: Glucocorticoid: 0.5-1.0 mg/kg/d prednisone (or other glucocorticoids of equivalent dose) for 1 month (visit V2-V3), then reduced by 5 mg every 2 weeks, and maintained at 5-10 mg/day to visit V8.
  Cyclophosphamide: intravenous infusion, once a month, 0.5-1g/m2 each time, 6 times in total, until the end of visit V7.
  Interventions: Drug: tofacitinib
- Glucocorticoids combined with tofacitinib Group: Glucocorticoid: 0.5-1.0 mg/kg/d prednisone (or other glucocorticoids of equivalent dose) for 1 month (visit V2-V3), then reduced by 5 mg every 2 weeks, and maintained at 5-10 mg/day to visit V8.
  Tofacitinib: oral, twice a day, 5mg each time, lasting for 6 months, until the end of visit V8.
  Interventions: Drug: tofacitinib

INTERVENTIONS:
Drug: tofacitinib — All subjects were treated immediately after non randomized enrollment. The treatment scheme of the experimental group: glucocorticoid+tropitib; the treatment scheme of the control group: glucocorticoid+cyclophosphamide.
  Other Names: cyclophosphamide

SUMMARY:
Compared with cyclophosphamide, the efficacy and safety of tofacitinib in the treatment of active IgG4-related diseases were evaluated.

DETAILED DESCRIPTION:
This study is a prospective, single center, non randomized, controlled, open label clinical observation study to evaluate the efficacy and safety of tropitib versus cyclophosphamide in inducing remission in IgG4-RD patients.

2) Investigators observe the diagnosis and treatment of IgG4-RD patients, and only provide patients with clinically appropriate diagnosis and treatment proposals.

It does not interfere with the choice of treatment plan for patients with the study drug of tropib or cyclophosphamide. If the patient chooses the hormone combined with tofatib or the hormone combined with cyclophosphamide as the main treatment drug, and at the same time meets the inclusion and exclusion criteria of this study, the patient can be included in this clinical observation study and become a subject. The experimental group was treated with glucocorticoid combined with tofatib, and the control group was treated with glucocorticoid combined with cyclophosphamide. It is planned that 20 people in each group will be treated for 6 months. After the study, the number of subjects in each group shall be at least 20 according to the actual situation. In the final statistical analysis, ensure that the sample size of the two groups participating in the statistical analysis is controlled at about 1:1.

3) The primary end point of this study was to compare the remission rate of the two groups after treatment; The secondary end point was to compare the response rate, recurrence rate and adverse event rate of the two groups after treatment.

ELIGIBILITY:
Inclusion Criteria:

* It meets the 2019 ACR/EULAR classification diagnostic criteria for IgG4 related diseases, and is an active IgG4-RD, defined as an IgG4-RD RI score ≥ 3 points when screening

Exclusion Criteria:

* 1. IgG4 related diseases endangering organ function or life;

  2. Only Mikulicz disease, no other internal organs involved;

  3. People with history of thrombotic disease or high risk of thrombosis;

  4. Have a history of malignant tumor;

  5. Active infection;

  6. Pregnant or lactating women;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IgG4-RD
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease remission rate at 1 month, 3 months and 6 months of treatment (%) | 1 month, 3 months and 6 months of treatment
  Definition of disease remission: including ① complete remission (CR) (main efficacy index), partial remission (PR), continuous complete remission (CCR) and no change (NC).

SECONDARY OUTCOMES:
Response rate at 1 month, 3 months and 6 months after treatment (%) | 1 month, 3 months and 6 months after treatment
  Defined as IgG4-RD RI score decrease ≥ 1 point
Disease recurrence rate at 3 and 6 months after treatment (%) | 3 and 6 months after treatment
  There are two types of disease recurrence, clinical recurrence and serological recurrence. Clinical recurrence was defined as recurrence of clinical symptoms or deterioration of imaging findings, with or without elevated serum IgG4 levels; Serological relapse was defined as an increase in serum IgG4 level and an increase in IgG4-RD RI score of ≥ 1 point after treatment, without recurrence of clinical symptoms or deterioration of imaging manifestations. The isolated increase of serum IgG4 concentration only constitutes serological recurrence. The date of recurrence is the date of onset of symptoms, or the date of new or deteriorated physical examination, laboratory examination or radiological examination results.
Changes in physician's overall assessment (PGA) from baseline at 1 month, 3 months and 6 months of treatment | 1 month, 3 months and 6 months of treatment
  First, the doctor evaluated the overall situation of IgG4 - RD subjects and marked them at the corresponding position of the straight line in the form of a vertical vertical line "l". The straight line is a 100mm scale, where the 0 end of the straight line represents very good, and the 100mm end represents very poor.

OTHER OUTCOMES:
Changes in the number of organs involved and IgG4-RD RI scores from the baseline after 6 months of treatment | 6 months of treatment
  The IgG4-RD RI value is obtained by superimposing the individual organ/site score of the patient. The score range of each organ/part is 0-3 points, which is defined as follows: 0 point means that the organ/part is not involved or completely relieved; 1: The lesions improved but still existed; 2 points: (after drug withdrawal) there was a new disease or recurrence of the previously involved site, or the disease did not improve after treatment; 3 Divided into (despite treatment) deterioration of lesions or new lesions.
  *When the disease of an important affected organ is urgent and requires active treatment, the score of the organ shall be doubled.
Changes of IgG4 level and related immunological indicators from baseline after 6 months of treatment | 6 months of treatment
  Relevant immune indicators include erythrocyte sedimentation rate, CRP, immunoglobulin, complement, IgG4, ANA spectrum, RF, ANCA, lymphocyte subsets, and cellular factor

CONTACTS AND LOCATIONS:
Overall Officials: Gao Jie, doctor, Study Chair — Changhai Hospital
Locations (1):
- Shanghai Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No